CLINICAL TRIAL: NCT01305317
Title: Study of Statins' Effect on Serum IgG, IgA Ang IgM Level in Chronic Hemodialysis Patients
Brief Title: Effect of Statins on IgG, IgA and IgM Level in Chronic Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Hamidreza Mahboobi, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: statins and Immunoglobulins
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2006-01

CONDITIONS: Chronic Kidney Disease
Keywords: Statin
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- lipitor (Experimental): atorvastatin 20mg daily
  Interventions: Drug: Lipitor

INTERVENTIONS:
Drug: Lipitor — Atorvastatin 20mg daily for 6 months
  Other Names: atorvastatin, statins

SUMMARY:
This is double blind randomized controlled trial on the statins effects on serum IgG, IgA and IgM level in chronic hemodialysis patients in Bandarabbas

DETAILED DESCRIPTION:
This study is a randomized controlled trial of statins effect on serum IgG, IgA and IgM level on chronic hemodialysis patients in Bandarabbas. The study is carried out in Hormozgan, Iran. Seventy four patient were randomized either to receive atorvastatin in addition of usual treatment or not. The primary outcomes were serum IgG,IgA and IgM level. The secondary outcome was drug side effects.

ELIGIBILITY:
Inclusion Criteria:

* All chronic hemodialysis patients attending Shahid Mohammadi hospital during the study period
* Accepting to participate in the study

Exclusion Criteria:

* Refusing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Serum IgG, IgA and IgM level | 6 months

SECONDARY OUTCOMES:
Drug side effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamidreza Mahboobi, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Shahid Mohammadi hospital, Bandar Abbas, Hormozgan, Iran